CLINICAL TRIAL: NCT03835637
Title: A Phase 1 Study of the Oral Glucocorticoid Receptor (GR) Antagonist ORIC-101 in Adult Healthy Subjects
Brief Title: Single and Multiple Dose Study of ORIC-101 in Adult Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ORIC-GR-17002
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Regimen A (Experimental)
  Interventions: Drug: ORIC-101
- Regimen B (Experimental)
  Interventions: Drug: ORIC-101
- Regimen C (Experimental)
  Interventions: Drug: ORIC-101
- Regimen D (Experimental)
  Interventions: Drug: ORIC-101
- Regimen F (Experimental)
  Interventions: Drug: ORIC-101
- Regimen H (Experimental)
  Interventions: Drug: ORIC-101
- Regimen I (Experimental)
  Interventions: Drug: ORIC-101

INTERVENTIONS:
Drug: ORIC-101 — Capsule or oral suspension

SUMMARY:
This is a single centre, open-label, non-randomised study with up to 2 parts, assessing the safety, tolerability, PK and PD of single (Part A) and multiple (Part B; optional) doses of oral GR antagonist ORIC-101.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-child bearing potential
* Age 18 to 65 years of age
* Body mass index of 18.0 to 32.0 kg/m^2 and weight between 50 kg and 120 kg, inclusive

Exclusion Criteria:

* Subjects who have received any investigational medicinal product (IMP) in a clinical research study within the previous 3 months
* History of any drug or alcohol abuse in the past 2 years
* Current smokers and those who have smoked within the last 12 months
* Females of childbearing potential
* Women with a history of unexplained vaginal bleeding or endometrial hyperplasia with atypia or endometrial carcinoma
* Current disease requiring treatment with systemic corticosteroids
* Serious adverse reaction or serious hypersensitivity to mifepristone, or any other drug, or the formulation excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 96 hours post-final dose
  PK of ORIC-101 as single doses
Area under the curve (AUC) | 96 hours post-final dose
  PK of ORIC-101 as single doses
Number of participants with adverse events | 96 hours post-final dose
  Safety and tolerability of ORIC-101 as single doses
Number of Participants With Abnormal Laboratory Values | 96 hours post-final dose
  Safety and tolerability of ORIC-101 as single doses

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 96 hours post-final dose
  Comparison of the PK of ORIC-101 in the presence or absence of food
Area under the curve (AUC) | 96 hours post-final dose
  Comparison of the PK of ORIC-101 in the presence or absence of food
Number of participants with adverse events | 96 hours post-final dose
  Safety and tolerability of ORIC-101 as multiple doses
Number of Participants With Abnormal Laboratory Values | 96 hours post-final dose
  Safety and tolerability of ORIC-101 as multiple doses
Maximum plasma concentration (Cmax) | 96 hours post-final dose
  PK of ORIC-101 as multiple doses
Area under the curve (AUC) | 96 hours post-final dose
  PK of ORIC-101 as multiple doses

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center, Nottingham, United Kingdom